CLINICAL TRIAL: NCT04972461
Title: Evaluate the Therapeutic Response by Using in Vitro Circulating Tumor Cell Expansion System
Brief Title: Therapeutic Response Evaluation by CTC Expansion System
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N201803020
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Circulating Tumor Cells
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Expanded circulating tumor cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among biomarkers, CTCs are a convenient, sensitive and biologically informative option. CTC detection could be considered a real-time "liquid biopsy" approach and contains several advantages such as minimally invasive, easy and safe to perform, and multiple samples can be taken over time, better prognosis to indicate an elevated risk of metastases, improved therapy monitoring, providing live disease status information., However, the number of CTCs is very low, so the establishment of cell culture from CTCs becomes the most challenging over the past year. In this study, we develop a short-term CTC expansion protocol combined with a new surface coating technique. Expanded circulating tumor cells will provide genetic information and develop oncology drug screening platform, which provides an opportunity to monitor response to therapy noninvasively.

DETAILED DESCRIPTION:
CTC detection could be considered a real-time "liquid biopsy" approach and contains several advantages such as minimally invasive, easy and safe to perform, and multiple samples can be taken over time, better prognosis to indicate an elevated risk of metastases, improved therapy monitoring, providing live disease status information., However, the number of CTCs is very low so the establishment of cell culture from CTCs becomes the most challenging over the past year. In this proposal we will develop a short-term CTC expansion protocol through combine with a new type of surface coating technique. Expanded circulating tumor cells will provide genetic information and develop oncology drug screening platform which provide an opportunity to noninvasively monitor response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant tumors

Exclusion Criteria:

* Unsuitable for recruitment by clinical judgement or non-compliance with regular follow-up.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced or metastatic solid tumors were enrolled. Eligible patients were ≥ 20 years old and had a life expectancy of more than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2023-08-07 (Estimated)

PRIMARY OUTCOMES:
To correlate drug sensitivity profiles of the expanded circulating tumor cells with the clinical treatment response. | CTC was expanded in vitro and drug sensitivity profile to disease-specific panels was obtained. The patient continued with the planned treatment by the treating physician and follow up information was obtained 3 months after blood sampling.
  CTC was expanded in vitro culture system and drug sensitivity profile to disease-specific panels was obtained. Clinical treatment response and drug sensitivity profile were analysed with 2 by 2 contingency tables. The evaluation of clinical response rate used by Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. Briefly, C+ refers to patients with clinical disease control (complete response, partial response, and stable disease), and C- refers to patients were found with worsening diseases (PD). Patients that did not fit into either category were listed as non-evaluable. The drug sensitivity profiles were categorized into E+ and E-. In class E+, at least one chemical in the evaluable treatment regimen was found to kill more than 30% of the cells in the CTC culture system. In class E-, all chemicals in the evaluable treatment regimen were found to kill less than 30% of the cells in the CTC culture system.

CONTACTS AND LOCATIONS:
Overall Officials: Long-Sheng Lu, MD, Ph.D., Study Director — Taipei Medical University Hospital; Jeng-Fong Chiou, MD, Ph.D., Study Chair — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantel K, Brakenhoff RH, Brandt B. Detection, clinical relevance and specific biological properties of disseminating tumour cells. Nat Rev Cancer. 2008 May;8(5):329-40. doi: 10.1038/nrc2375. PMID 18404148
- [Background] Muller V, Riethdorf S, Rack B, Janni W, Fasching PA, Solomayer E, Aktas B, Kasimir-Bauer S, Pantel K, Fehm T; DETECT study group. Prognostic impact of circulating tumor cells assessed with the CellSearch System and AdnaTest Breast in metastatic breast cancer patients: the DETECT study. Breast Cancer Res. 2012 Aug 15;14(4):R118. doi: 10.1186/bcr3243. PMID 22894854
- [Derived] Wu YH, Chao HS, Chiang CL, Luo YH, Chiu CH, Yen SH, Liu CY, Chiou JF, Burnouf T, Chen YJ, Wang PY, Chao TY, Hsu SM, Lu LS. Personalized cancer avatars for patients with thymic malignancies: A pilot study with circulating tumor cell-derived organoids. Thorac Cancer. 2023 Sep;14(25):2591-2600. doi: 10.1111/1759-7714.15039. Epub 2023 Jul 20. PMID 37474689

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04972461/Prot_ICF_000.pdf